CLINICAL TRIAL: NCT03993080
Title: Virtual Reality Relaxation to Decrease Dental Anxiety in Primary Dental Care
Brief Title: Virtual Reality Relaxation to Decrease Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of St Andrews (Other); University of Dundee (Other); City of Helsinki (Other)
Responsible Party: Principal Investigator, Satu Lahti, Professor of Community Dentistry, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEL 2018-008940
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; virtual reality

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-center trial with two parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality relaxation (Experimental): Virtual reality relaxation using virtual landscape and audio features and sound
  Interventions: Device: Virtual reality relaxation
- Treatment as usual (No Intervention): Seated in similar environment as experimental group for same time

INTERVENTIONS:
Device: Virtual reality relaxation — 1-3.5 minute 360° videos
  Arms: Virtual reality relaxation

SUMMARY:
The aim is to apply short-term virtual reality relaxation to examine if it is effective in reducing pre-operative dental anxiety in primary health care using an RCT.

DETAILED DESCRIPTION:
Randomized controlled single-center trial with two parallel arms: Virtual Reality Relaxation (VRR) and Treatment As Usual (TAU) in a public oral health care unit. VRR group receiving a 1-3.5 minute 360° video immersing them in peaceful virtual landscape with audio features and sound supporting the relaxing experience. TAU groups remaining seated for 3 minutes in similar setting.

ELIGIBILITY:
Inclusion Criteria:

* attending for dental treatment
* consenting
* able to complete Finnish questionnaire without assistance
* age 18 years or older

Exclusion Criteria:

* those not meeting inclusion criteria

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Dental anxiety | immediately after intervention
  post-test measured with Modified Dental Anxiety Scale, The measure has five questions, each with five reply alternatives from not anxious to extremely anxious (on a scale 1-5), MDAS sums up to the total scale (range 5-25) which is used as primary outcome. Higher scores indicate higher dental anxiety.

SECONDARY OUTCOMES:
Anticipatory dental anxiety and treatment related dental anxiety | immediately after intervention
  The secondary outcome variables are post-test scores for the two sub-scales of the MDAS referred to as 'anticipatory' (MDAS items 1 and 2) and 'treatment' dental anxiety (MDAS items 3, 4 and 5). Scales for sum up as anticipatory anxiety (Items 1 and 2: range 2-10) and treatment anxiety (Items 3-5, range 3-15). Higher scores indicate higher dental anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Satu Lahti, Principal Investigator — Department of Community Dentistry, University of Turku, Finland
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lahti S, Suominen A, Freeman R, Lahteenoja T, Humphris G. Virtual Reality Relaxation to Decrease Dental Anxiety: Immediate Effect Randomized Clinical Trial. JDR Clin Trans Res. 2020 Oct;5(4):312-318. doi: 10.1177/2380084420901679. Epub 2020 Jan 21. PMID 31962052